CLINICAL TRIAL: NCT05046951
Title: Testing Methods to Increase Lung Cancer Screening Among Quitline Callers
Brief Title: Educating QUitline Callers About Lung Cancer Screening
Acronym: EQUAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00002708
Record Dates: First submitted 2021-06-08; First posted 2021-09-16 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Population at Risk
Keywords: lung cancer; lung cancer screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web arm (Active Comparator): The Should I Screen educational website, developed by our consultant, Rafael Meza, PhD, is available at no cost, is written at an 8th grade reading level, requires 15 minutes to use, and undergoes regular updates (https://shouldiscreen.com). The goal is to increase lung screening awareness and to encourage a shared decision making visit with a provider. Sections of the website include the benefits (the reduced likelihood of dying from lung cancer) and harms (false alarms, overdiagnosis, more testing, and invasive procedures) of screening, causes of lung cancer, methods to reduce lung cancer risk, and the lung cancer risk calculator. Improvements in knowledge have been demonstrated with individuals eligible for screening.
  Interventions: Behavioral: Should I Screen website
- Print Arm (Active Comparator): The Should I Screen print-based education (included with this IRB protocol) will be developed in Aim 1 and compared to the Should I Screen website in Aim 2. It will also be at the 8th grade level and will require 15 minutes to read. Although it will contain the same topics as the website, there is one inherent difference - it is not possible to include the interactive risk calculator in the print version. The print-based version will list all of the risk criteria that are included in the algorithm so that participants can see which ones apply to them. However, the risk calculator requires the computer algorithm to calculate a person's 6-year risk of developing lung cancer.
  Interventions: Behavioral: Should I Screen print booklet

INTERVENTIONS:
Behavioral: Should I Screen website — The Should I Screen educational website, developed by our consultant, Rafael Meza, PhD, is available at no cost, is written at an 8th grade reading level, requires 15 minutes to use, and undergoes regular updates (https://shouldiscreen.com). The goal is to increase lung screening awareness and to encourage a shared decision making visit with a provider. Sections of the website include the benefits (the reduced likelihood of dying from lung cancer) and harms (false alarms, overdiagnosis, more testing, and invasive procedures) of screening, causes of lung cancer, methods to reduce lung cancer risk, and the lung cancer risk calculator. Improvements in knowledge have been demonstrated with individuals eligible for screening.
  Arms: Web arm
Behavioral: Should I Screen print booklet — The Should I Screen print-based education will be developed in Aim 1 and compared to the Should I Screen website in Aim 2. It will also be at the 8th grade level and will require 15 minutes to read. Although it will contain the same topics as the website, there is one inherent difference - it is not possible to include the interactive risk calculator in the print version. The print-based version will list all of the risk criteria that are included in the algorithm so that participants can see which ones apply to them. However, the risk calculator requires the computer algorithm to calculate a person's 6-year risk of developing lung cancer.
  Arms: Print Arm

SUMMARY:
The specific aims are:

1. To evaluate the potential barriers of providing educational lung screening interventions to quitline users, the investigators will seek input from 10-20 stakeholders on the newly adapted print version of the Should I Screen website, and on our proposed Aim 2 recruitment and retention procedures.
2. To conduct a randomized intervention, comparing: 1) ShouldIScreen.com website, (WEB; N=150); vs. 2) the Should I Screen print version (PRINT; N=150). H2.1. At 1- and 4-months post-randomization, the WEB arm will have significantly higher lung screening knowledge and intention to undergo lung screening, compared to PRINT. Randomization will be stratified by age and pack-years in order to incorporate those who are recently eligible for screening, ages 50-54 and with 20-29 pack years. H2.2 The investigators will explore several potential moderators (age and e-health literacy). For example, the investigators will explore whether older vs younger participants have differential knowledge outcomes when using the PRINT vs WEB interventions. H2.3 We will explore whether mediators (prior lung screening, current primary care provider, lung cancer perceived risk) positively affects knowledge and screening intentions.
3. To evaluate reach (% of quitline users enrolled) and engagement (% who read the intervention materials) by study arm and subgroup (e.g., method of quitline access, age, e-health literacy).

DETAILED DESCRIPTION:
Aim 1: The 30-45 minute qualitative interviews will obtain: 1) feedback on the print adaptation of the Should I Screen website (the investigators will send it in advance of the interview), 2) recommendations for effective recruitment and retention procedures in Aim 2, 3) feedback on methods to increase the likelihood that participants will enroll and engage with the interventions (e.g., whether to present the study information immediately following initial contact with the quitline or later), 4) ideas to increase the likelihood that participants will contact their providers for an appointment to discuss lung screening, and 5) feedback on the Aim 2 measures regarding feasibility and acceptability.

Aim 2: H2.1. At 1- and 4-months post-randomization, the WEB arm will have significantly higher lung screening knowledge and intentions to undergo lung screening, compared to PRINT. H2.2 Moderators include, age, e-health literacy. For example, the investigators expect that younger participants will have significantly increased knowledge in the WEB (vs PRINT) arm, whereas intervention arm will have less of an impact among the older participants. H2.3 Mediators (e.g., prior lung screening, current primary care provider, lung cancer perceived risk) will positively affect knowledge and screening intentions. Aim 3. To evaluate reach (% of quitline users enrolled) and engagement (% who read the intervention materials) by study arm and subgroup (e.g., age, e-health literacy). The investigators will assess the feasibility for widespread implementation of both interventions

ELIGIBILITY:
Inclusion Criteria:

* enrolled in the quitline
* 50-80 years old
* >20-pack year smoking history
* never screened or >12 months since prior screen
* English speaking
* able to provide meaningful consent
* no family members in the same household enrolled in the trial

Exclusion Criterion:

* prior lung cancer

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Reach of eligible quitline users | baseline assessment
  % of eligible quitline users enrolled in the trial;
Intervention Engagement of eligible quitline users | one month assessment
  WEB: electronic assessment of 1) logged on, 2) total time spent on website, 3) sections accessed; PRINT: self-reported time spent reading;
Satisfaction with the intervention materials. | one month assessment
  Assessment of satisfaction with length, format, and content of the materials
Lung cancer screening knowledge | one month assessment
  Assessment of lung cancer risk factors, screening eligibility, and pros/cons of screening
Lung cancer screening knowledge | four month assessment
  Assessment of lung cancer risk factors, screening eligibility, and pros/cons of screening
Percentage of participants who intend to undergo lung cancer screening | one month assessment
  Intent to undergo lung cancer screening
Percentage of participants who intend to undergo lung cancer screening | four month assessment
  Intent to undergo lung cancer screening

SECONDARY OUTCOMES:
Percentage of participants with an appointment for a shared decision making visit | one month assessment
  Shared decision making appt, lung screening referral, completed lung scan.
Percentage of participants with an appointment for a shared decision making visit | four month assessment
  Shared decision making appt, lung screening referral, completed lung scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers can email the corresponding author to request access to deidentified data. A data analyais plan and IRB approval will be required.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be availble for one year following the date of publication.
Access Criteria: Email the corresponding author with the request. Kathryn L. Taylor, taylorkl@georgetown.edu

REFERENCES:
- [Background] Webster M, Whealan J, Williams RM, Eyestone E, Le A, Childs J, Kao JY, Martin M, Wolfe S, Yang F, Hung PY, Lau YK, Luta G, Tammemagi M, Meza R, Taylor KL. The tobacco quitline setting as a teachable moment: The Educating Quitline Users About Lung (EQUAL) cancer screening randomized trial. Transl Behav Med. 2023 Sep 28;13(10):736-747. doi: 10.1093/tbm/ibad049. PMID 37616531